CLINICAL TRIAL: NCT00001627
Title: Collection of Blood and Bone Marrow From Healthy Volunteers and Patients for Research Purposes
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970130; 97-H-0130
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Bone Marrow Diseases; Healthy Volunteers
Keywords: Bone Marrow; Hematopoiesis; DNA; RNA; Viruses
MeSH Terms: conditions — Bone Marrow Diseases; Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group 1: Normal Volunteers and patients.

SUMMARY:
This study is designed to provide bone marrow and/or blood cells for other research studies. Patients participating in this study will be asked to provide small amounts of medical information and undergo a limited physical examination designed to detect the presence of any obvious blood disease. A blood and bone marrow sample will be obtained to verify that the patient has normal blood cell production.

Researchers plan to obtain bone marrow samples to be used in laboratory studies directed toward understanding the formation of blood cells. Bone marrow samples will be taken from the hip bone of patients and healthy volunteers.

These samples are valuable to many research studies within the Hematology Branch of the National Heart, Lung, and Blood Institute, including studies of normal and abnormal production of blood cells, the viral causes of blood diseases, and the role of the immune system in bone marrow failure and related conditions....

DETAILED DESCRIPTION:
This protocol defines in general terms the purposes for which blood and bone marrow specimens will be collected by members of the Hematology Branch and the conditions under which the sampling will be performed. Samples of blood and bone marrow from healthy volunteers and from patients are indispensable for many research projects, including studies of normal and abnormal hematopoiesis, the viral etiology of blood diseases, and the role of the immune system in marrow failure and related conditions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers age greater than or equal to 18 years.

Subjects with hematologic disease age greater than or equal to 2 (for subjects less than 18, blood and bone marrow specimens will be obtained concurrently with clinically indicated sampling).

EXCLUSION CRITERIA:

History of a significant bleeding disorder.

Abnormal host-defense mechanisms.

Ages: 2 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Normal Volunteers and patients
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 1997-07-08 (Actual); Primary Completion 2010-12-22 (Actual); Study Completion 2010-12-22 (Actual)

PRIMARY OUTCOMES:
To provide a readily available supply of samples for blood and bone marrow for in vitro studies in the Hematology Branch laboratories | Ongoing
  The collection of adequate cells for laboratory research.

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-H-0130.html